CLINICAL TRIAL: NCT06804902
Title: Improving the Accuracy of Malaria RDT Reporting in Public Primary Healthcare Facilities in Côte d'Ivoire
Brief Title: MaCRA Part B in Côte d'Ivoire
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: USAID termination of project funding and activities
Sponsor: PATH (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Institut National de Sante Publique (Other); US President's Malaria Initiative (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RES-00849
Record Dates: First submitted 2025-01-22; First posted 2025-02-03 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Health facilities in intervention districts will bring all RDT cassettes performed in their facility and all outpatient registers to a monthly data validation meeting led by the surveillance, monitoring and evaluation officers (CSE). During these meetings, Audere's HealthPulse application will be used to take photos of each facility's RDT cassettes, tallying the total number of RDTs and total by result. The test positivity rates (TPRs) from the registers will be manually entered into the application and compared with the TPR from the RDT photos. Healthcare facilities with a discrepancy above a certain threshold between TPR derived from register data and the TPR derived from the RDT images may be asked to carry out a more detailed audit to better understand the source of discrepant results. If discrepancies are identified, the CSE will determine what corrections are required before entry into the DHIS2.
  Interventions: Behavioral: Monthly RDT Validation Meeting
- Control (No Intervention): There will be no activities in the control arm.

INTERVENTIONS:
Behavioral: Monthly RDT Validation Meeting — Health facilities in intervention districts will bring all RDT cassettes performed in their facility and all outpatient registers to a monthly data validation meeting led by the surveillance, monitoring and evaluation officers (CSE). During these meetings, Audere's HealthPulse application will be used to take photos of each facility's RDT cassettes, tallying the total number of RDTs and total by result. The test positivity rates (TPRs) from the registers will be manually entered into the application and compared with the TPR from the RDT photos. Healthcare facilities with a discrepancy above a certain threshold between TPR derived from register data and the TPR derived from the RDT images may be asked to carry out a more detailed audit to better understand the source of discrepant results. If discrepancies are identified, the CSE will determine what corrections are required before entry into the DHIS2.
  Arms: Intervention

SUMMARY:
This study aims to evaluate the effectiveness of monthly malaria rapid diagnostic test (RDT) validation meetings at district level on reducing the proportion of RDT results recorded as positive in health facility registers in Cote d'Ivoire.

DETAILED DESCRIPTION:
PMI Insights supported a multi-country evaluation of the accuracy of the recording and reporting of rapid diagnostic test (RDT) results at health facilities in Benin, Côte d'Ivoire, Nigeria, and Uganda (MaCRA Part A). The evaluation found a high degree of agreement between RDT results recorded in health facilities and an objective panel reading of the same RDTs. However, the changes in test positivity rate (TPR) after the start of the study suggest that some of this agreement may have been a result of the Hawthorne effect: in all countries except Benin, TPR declined after the start of the evaluation in facilities where evaluation staff were present, compared with control facilities. This suggests that the presence of evaluation staff caused health care workers to change their behavior with respect to reporting positive RDT results. The study evaluated the durability of RDT results and found that 95% of RDT cassettes retained their original reading over a one-month period. This provides evidence that stored RDT cassettes may be compared to health facility registers at monthly validation meetings, as long as a certain margin of error is used to account for the proportion of tests that may change.

The results from the first phase of the study were used to identify potential interventions to improve RDT reporting and recording accuracy in health facilities. The second phase of the study aims to evaluate the effectiveness of monthly district-level RDT result validation meetings on reducing the proportion of RDT results recorded as positive in health facility registers and reported to the national health management information system.

This is a two-arm cluster-randomized controlled effectiveness evaluation. Districts will serve as the clusters and will be assigned using restricted randomization to the intervention or control arm. In the intervention arm, the Ministry of Health will lead monthly district-level RDT validation meetings facilitated by a digital phone-based app which uses AI to record RDT results (HealthPulse, Audere, Johannesburg, South Africa). There will be no study activities in the control facilities.

Monthly RDT validation meetings will take place over a four-month period (April to July 2025), after which a cross-sectional survey and in- depth interviews will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers responsible for testing or interpreting malaria RDTs in the selected study facilities
* District and regional health teams involved in the monthly RDT validation meetings from districts selected for the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The proportion of RDTs recorded as positive in healthcare facility registers. | Four months
  Data will be collected from the DHIS2 after the end of the study for both control and intervention arms.

SECONDARY OUTCOMES:
Ratio of TPR between healthcare facility registers and RDT cassettes in intervention facilities over time. | Four months
  The TPR for RDT cassettes will be collected from each healthcare facility by the HealthPulse application during monthly RDT validation meetings. The ratio will be calculated with these data, and the TPRs calculated from DHIS2.
Proportion of suspected patients tested by RDT who receive an antimalarial prescription. | Four months
  For both the intervention and control arms, data on ACT prescription will be downloaded from the DHIS2 after the end of the study.
The total number of antimalarials. | Four months
  For both arms, ACT prescription data will be downloaded from the DHIS2, and ACT consumption data from the integrated electronic logistics management system (e-SIGL) after the end of the study.
The cost required to implement the monthly RDT validation meetings. | Four months
  This estimate will be made by recording the cost of training, the cost of smartphones and communication time, the number and categories of staff needed to plan and implement the monthly data validation meetings, as well as their travel expenses and per diems for attending the meeting. The costs of any follow-up activities will be noted. The time spent by different categories of staff will be tracked to provide an estimate of the level of effort required to implement the monthly validation meetings.
Proportion of healthcare workers reporting compliance with negative RDT results when patients present with fever (i.e. recording the RDT result as negative, not recording the case as malaria and not prescribing antimalarial medication). | immediately after the intervention period
  Subjective norms, attitudes and practices towards RDTs will be measured in a cross-sectional survey of healthcare workers in selected facilities at the end of the study.
Qualitative description of the acceptability and feasibility of conducting monthly RDT validations and using a digital tool (HealthPulse, Audere, Johannesburg, South Africa). | immediately after the intervention period
  The acceptability and feasibility of the monthly RDT validation exercise, as well as perceptions of the digital tools used for RDT validation, will be measured through in-depth interviews with health facility staff, district epidemiological surveillance and monitoring and evaluation (CSE) officers and malaria focal points.

CONTACTS AND LOCATIONS:
Overall Officials: William Yavo, Principal Investigator — INSP
Locations (1):
- Health facilities in selected districts, Cities in Selected Districts, Côte d’Ivoire